CLINICAL TRIAL: NCT01496417
Title: A 12 Month, Single-center, Non-randomized, Open-label Study of Outcomes of Intermediate Risk Maryland Aggregate Pathology Index (MAPI) Scores in de Novo Renal Transplant Recipients
Brief Title: Belatacept in Renal Transplantation With Intermediate Risk Maryland Aggregate Pathology Index (MAPI) Scores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Rolf Barth, Principal Investigator, University of Maryland
Organization: University of Maryland, Baltimore (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP00048573
Record Dates: First submitted 2011-12-14; First posted 2011-12-21 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: End-Stage Renal Disease
Keywords: Kidney Transplantation; Biopsy; Belatacept
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belatacept therapy (Experimental): 20 Patients receiving belatacept based immunosuppressive protocol for 12 months post-transplantation.
  Interventions: Drug: Belatacept

INTERVENTIONS:
Drug: Belatacept — Belatacept infusion intravenous at 10 mg/kg on post-operative days 1, 5, and weeks 2, 4, 8, 12; 5mg/kg intravenous dose at weeks 16, 20, 24, 28, 32, 36, 40, 44, and 48.
  Other Names: Nulojix

SUMMARY:
This will be a pilot study to investigate the use of belatacept (BMS) therapy in kidney transplant patients who have a MAPI score of greater than or equal to 8. The MAPI (Maryland Aggregate Pathology Index) score is a preimplantation donor scoring system which has five histopathological parameters that impact long-term kidney outcomes. Many kidney transplant recipients use calcineurin inhibitors (CNIs) as one of their anti-rejection medi cations. Kidney function may be affected by anti-rejection medications known as calcineurin inhibitors (CNIs). Sometimes CNIs can lead to toxicities and eventually loss of the kidney or episodes of chronic allograft nephropathy (CAN). Avoiding CNI immunosuppression and using belatacept therapy (BMS) instead, may be associated with improved kidney transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female renal recipients 18-70 years of age undergoing primary kidney transplantation.
* Recipients of deceased donor (including expanded criteria donor organs and deceased donor organs after cardiac death) with MAPI score ≥ 8.
* Cold ischemic time less than 40 hours at time of reperfusion.
* Negative serum pregnancy test for female patients.
* Patients who can understand the purposes and risks of the study, provide informed consent, and can comply with the treatment and follow-up requirements.

Exclusion Criteria:

* Cold ischemic time (CIT) > 40 hours
* Patients who are sensitized with current PRA>40%, ABO incompatible transplants, or T, or B cell crossmatch positive transplant.
* Patients without antibody to EBV
* Patients receiving multiple organ transplants.
* Patients unable to take oral medication at time of randomization
* Patient with a history of malignancy of any organ system, treated or untreated, within the past 2 years whether or not there is evidence of local recurrence or metastases, with the exception of carcinoma in situ
* Patients who tested positive for HIV, Hepatitis C or Hepatitis B surface antigen.
* Recipients of organs from donors who test positive for HIV, Hepatitis C or Hepatitis B surface antigen
* Patients with a clinically significant systemic infection within 30 days prior to transplant
* Patients who have cardiac failure at time of screening or any other severe cardiac disease as determined by the investigator
* Patients with abnormal laboratory findings of clinical significance within 2 weeks of randomization which would interfere with the objectives of the study.
* Females, pregnant or lactating, or are of childbearing potential unwilling to use an effective means of contraception or are planning to become pregnant.
* Patient with active tuberculosis infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2017-02-28 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Renal Function | 12 months
  To evaluate renal function in Belatacept treated recipients of intermediate risk MAPI score allografts in terms of estimated glomerular filtration rate (eGFR, calculated using the MDRD formula) assessed at 12 months. The 12 month eGFR will be compared to existing cohorts of calcineurin inhibitor treated patients with MAPI scores above 8.

SECONDARY OUTCOMES:
Rejection rate | 12 months
  Secondary objectives include the biopsy proven rejection rates at 12 months and comparison to existing cohorts of calcineurin inhibitor treated patients.
Graft survival | 12 months
  Secondary objectives include renal allograft survival at 12 months.
MAPI biopsy score | 12 months
  Secondary objectives include the MAPI score at 3 and 12 months. The MAPI score change compared to baseline in the study group will be important in comparison to existing cohorts of calcineurin inhibitor treated patients, to determine whether calcineurin free-regimens are associated with both functional and histologic differences as compared to calcineurin based therapies.
Patient survival | 12 months
  Secondary objectives include patient survival at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf N Barth, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Background] Vincenti F, Blancho G, Durrbach A, Friend P, Grinyo J, Halloran PF, Klempnauer J, Lang P, Larsen CP, Muhlbacher F, Nashan B, Soulillou JP, Vanrenterghem Y, Wekerle T, Agarwal M, Gujrathi S, Shen J, Shi R, Townsend R, Charpentier B. Five-year safety and efficacy of belatacept in renal transplantation. J Am Soc Nephrol. 2010 Sep;21(9):1587-96. doi: 10.1681/ASN.2009111109. Epub 2010 Jul 15. PMID 20634298
- [Background] Vincenti F, Larsen C, Durrbach A, Wekerle T, Nashan B, Blancho G, Lang P, Grinyo J, Halloran PF, Solez K, Hagerty D, Levy E, Zhou W, Natarajan K, Charpentier B; Belatacept Study Group. Costimulation blockade with belatacept in renal transplantation. N Engl J Med. 2005 Aug 25;353(8):770-81. doi: 10.1056/NEJMoa050085. PMID 16120857
- [Background] Vincenti F, Charpentier B, Vanrenterghem Y, Rostaing L, Bresnahan B, Darji P, Massari P, Mondragon-Ramirez GA, Agarwal M, Di Russo G, Lin CS, Garg P, Larsen CP. A phase III study of belatacept-based immunosuppression regimens versus cyclosporine in renal transplant recipients (BENEFIT study). Am J Transplant. 2010 Mar;10(3):535-46. doi: 10.1111/j.1600-6143.2009.03005.x. PMID 20415897
- [Background] Larsen CP, Grinyo J, Medina-Pestana J, Vanrenterghem Y, Vincenti F, Breshahan B, Campistol JM, Florman S, Rial Mdel C, Kamar N, Block A, Di Russo G, Lin CS, Garg P, Charpentier B. Belatacept-based regimens versus a cyclosporine A-based regimen in kidney transplant recipients: 2-year results from the BENEFIT and BENEFIT-EXT studies. Transplantation. 2010 Dec 27;90(12):1528-35. doi: 10.1097/TP.0b013e3181ff87cd. PMID 21076381
- [Derived] Sparkes T, Ravichandran B, Opara O, Ugarte R, Drachenberg CB, Philosophe B, Bromberg JS, Barth RN. Alemtuzumab induction and belatacept maintenance in marginal pathology renal allografts. Clin Transplant. 2019 Jun;33(6):e13531. doi: 10.1111/ctr.13531. Epub 2019 Apr 11. PMID 30866104
- See also: University of Maryland Division of Transplantation — http://umm.edu/transplant